CLINICAL TRIAL: NCT05950347
Title: The Efficacy and Safety of Transcutaneous Auricular Vagus Nerve Stimulation for Anxiety in Parkinson's Disease
Brief Title: The Efficacy and Safety of Transcutaneous Auricular Vagus Nerve Stimulation for Anxiety in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Kezhong Zhang, professor，Chief physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-07
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Anxiety; taVNS
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Transcutaneous auricular vagus nerve stimulation (Active Comparator): Two modiﬁed dot-like electrodes delivered the stimulation to the cymba conchae of left ear in the vicinity of the auricular branch vagus nerve. Stimulation parameters: frequency = 20/4 Hz; pulse width = 200 μs; 20 Hz lasting 7 seconds, alternated with 4 Hz lasting 3 seconds，repeat until 30 min. Every PD patient received stimulation twice daily , 30 minutes each time, for 14 consecutive days. The stimulation intensity was set as the maximum value the patient could tolerate without causing pain.
  Interventions: Device: Active Transcutaneous auricular vagus nerve stimulation
- Sham Transcutaneous auricular vagus nerve stimulation (Sham Comparator): Two modiﬁed dot-like electrodes delivered the stimulation to the left earlobe. Stimulation parameters: frequency = 20/4 Hz; pulse width = 200 μs; 20 Hz lasting 7 seconds, alternated with 4 Hz lasting 3 seconds，repeat until 30 min. Every PD patient received stimulation twice daily , 30 minutes each time, for 14 consecutive days. The stimulation intensity was set as the maximum value the patient could tolerate without causing pain.
  Interventions: Device: Sham Transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: Active Transcutaneous auricular vagus nerve stimulation — Two modiﬁed dot-like electrodes delivered the stimulation to the cymba conchae of left ear in the vicinity of the auricular branch vagus nerve. Stimulation parameters: frequency = 20/4 Hz; pulse width = 200 μs; 20 Hz lasting 7 seconds, alternated with 4 Hz lasting 3 seconds，repeat until 30 min. Every PD patient received stimulation twice daily , 30 minutes each time, for 14 consecutive days. The stimulation intensity was set as the maximum value the patient could tolerate without causing pain.
  Arms: Active Transcutaneous auricular vagus nerve stimulation
Device: Sham Transcutaneous auricular vagus nerve stimulation — Two modiﬁed dot-like electrodes delivered the stimulation to the cymba conchae of left ear in the vicinity of the auricular branch vagus nerve. Stimulation parameters: frequency = 20/4 Hz; pulse width = 200 μs; 20 Hz lasting 7 seconds, alternated with 4 Hz lasting 3 seconds，repeat until 30 min. Every PD patient received stimulation twice daily , 30 minutes each time, for 14 consecutive days. The stimulation intensity was set as the maximum value the patient could tolerate without causing pain.
  Arms: Sham Transcutaneous auricular vagus nerve stimulation

SUMMARY:
This study is a double blind comparative study examining the effectiveness of the transcutaneous auricular vagus nerve stimulation treatment on Parkinson's disease patients with anxiety. The investigators hypothesize that taVNS will improve anxiety and cortical activity in Parkinson's disease patients with anxiety.

DETAILED DESCRIPTION:
Participants in the Experimental group underwent fourteen consecutive daily sessions of transcutaneous auricular vagus nerve stimulation (taVNS, twice daily, 30 minutes each time) , whereas participants in the sham stimulation group underwent fourteen consecutive daily sessions of sham taVNS. Assessments of anxiety symptoms, motor symptoms were performed three times: at baseline, one day post intervention and 2 weeks post intervention. The cortical activity (using Functional near-infrared spectroscopy) were assessed at baseline, one day post intervention.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosed with idiopathic PD according to the Movement Disorder Society Clinical Diagnostic Criteria for PD;
* (2) meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for anxiety and Hamilton Anxiety Scale (HAMA) score ≥ 12;
* (3) stable pharmacotherapy for PD at least one month prior to the study;
* (4) 40-80 years old;
* (5) willing to sign written informed consent.

Exclusion Criteria:

* (1) with cognitive impairment, according to Montreal Cognitive Assessment (MOCA) < 23;
* (2) took antianxiety drugs;
* (3) with taVNS contraindications;
* (4) received VNS treatment during the past month;
* (5) with concomitant severe neurologic, renal, cardiovascular, or hepatic disease.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
change of Hamilton Anxiety Scale Score | Assessed at baseline, one day post intervention，2 weeks post intervention
  Hamilton Anxiety Scale (HAM-A score), which was used for assessing the degree of anxiety. It consists of 14 symptomatic definition elements, with a total possible score of 56. The differences in HAMA score before and after treatment can be used to evaluate the effect of taVNS treatment.

SECONDARY OUTCOMES:
change of HbO2 in the prefrontal cortex | Assessed at baseline, one day post intervention
  The change of HbO2 in the prefrontal cortex is accessed by fNIRS combined with verbal fluency task. Recent documents have highlighted the effectiveness of fNIRS combined with verbal fluency task (VFT) in detecting alterations in the PFC in patients with anxiety. The differences in HbO2 before and after treatment can be used to evaluate the effect of taVNS treatment.
change of Uniﬁed Parkinson's Disease Rating Scale Score section III | Assessed at baseline, one day post intervention，2 weeks post intervention
  Uniﬁed Parkinson's Disease Rating Scale Score section III were used to assess the severity of motor symptoms.
change of Uniﬁed Parkinson's Disease Rating Scale Score section I | Assessed at baseline, one day post intervention，2 weeks post intervention
  Uniﬁed Parkinson's Disease Rating Scale Score section I can evaluate changes in mental state and cognition (including behavior and emotions)

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China